CLINICAL TRIAL: NCT07280091
Title: Study of Skin and Gut Microbiome in a Skin Condition Involving Skin Barrier Impairment and Allergic Symptoms: Netherton Syndrome
Acronym: DERMABIOTE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250480; ID-RCB Number (Other: 2025-A00300-49)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Netherton Syndrome
Keywords: Netherton syndrome; skin microbiome
MeSH Terms: conditions — Netherton Syndrome | interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Superficial skin swabs, Stool, Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Netherton syndrome: 15 children, adolescents, and young adults with Netherton syndrome
  Interventions: Biological: Superficial skin swabs; Biological: Stool samples; Biological: Saliva samples; Biological: Blood samples; Other: Data-Collection
- Control subjects: 15 control subjects of the same age group and gender, treated at the service but with no dermatosis or inflammatory and/or autoimmune diseases.
  Interventions: Biological: Superficial skin swabs; Biological: Stool samples; Biological: Saliva samples; Biological: Blood samples; Other: Data-Collection

INTERVENTIONS:
Biological: Superficial skin swabs — Sampling areas: (18 swabs in total + 6 swabs for routine skin mapping)
  1. Lesion area outside skin folds (e.g., back or limb)
  2. Healthy area outside skin folds (e.g., back or limb)
  3. Perioral area of the face
  4. Scalp
  5. Inguinal fold
  6. Axillary fold
  Groups: Patients with Netherton syndrome
Biological: Superficial skin swabs — Three superficial skin swabs: same locations as for Netherton patients
  Groups: Control subjects
Biological: Stool samples — A stool sample collected for analysis of the fecal microbiome and mycobiome.
Biological: Saliva samples — A saliva sample collected for analysis of the saliva microbiome and mycobiome.
Biological: Blood samples — For group A: cytokine profile from an additional blood sample taken during a blood draw for treatment For group B: cytokine profile if there is any residual blood sample from the treatment
  Groups: Control subjects
Biological: Blood samples — For group A: cytokine profile from an additional blood sample taken during a blood draw for treatment For group B: cytokine profile if there is any residual blood sample from the treatment
  Groups: Patients with Netherton syndrome
Other: Data-Collection — Socio-demographic data and lifestyle habits of the patient and parents
Other: Data-Collection — Clinical data, treatment data, and results of biological tests carried out as part of routine monitoring
  Groups: Patients with Netherton syndrome

SUMMARY:
It is proposed to conduct an exploratory study to analyze the skin, intestinal, and salivary microbiome, as well as the skin mycobiome and virome, of patients (adolescents and young adults) with Netherton syndrome, a condition characterized by an impaired skin barrier that most likely promotes the development of allergic manifestations.

The study will be conducted on patients with Netherton syndrome and control subjects in order to investigate possible correlation factors between the three microbiomes and identify which ones.

DETAILED DESCRIPTION:
Netherton syndrome (NS) is a genodermatosis characterized by the combination of (i) pruritic erythematous-squamous skin lesions, often erythrodermic, with inflammatory skin flare-ups, (ii) frequent hypernatremic dehydration in the neonatal period, (iii) food allergies with increased IgE levels, and (iv) growth retardation. Autosomal recessive in transmission, it is linked to mutations in the SPINK5 gene encoding the LEKTI protein, leading to abnormalities in epithelial barriers, particularly in the skin and esophagus. Digestive disorders such as abdominal pain, chronic diarrhea, or eosinophilic digestive disorders are common, as described by the dermatology team at Necker-Enfants Malades Hospital, MAGEC center. Thus, NS is a model of a rare disease combining skin inflammation and impaired epithelial barriers. It is essential to define all therapeutic strategies that can relieve patients of what is currently a chronic, severe, and orphan disease. Currently, there is no specific treatment available. The permeability of the skin barrier means that treatment with topical corticosteroids should be avoided as much as possible. Their use therefore remains very limited.

Recent data concerning the study of the skin microbiome of patients with SN have confirmed the presence of dysbiosis and shown the over-representation of Staphylococcus aureus and epidermidis strains, as well as the harmful role of certain proteases produced or stimulated by these strains. However, these studies involved a limited number of patients (a maximum of 10 NS patients), all adults, and did not include skin sampling sites of particular interest, such as skin folds in patients with chronic vegetative cellulitis, which is rarely described but observed in some NS patients. Furthermore, although these patients frequently present with digestive disorders, the digestive microbiome has never been studied in NS. A comparison between studies of the skin and digestive microbiome in systemic inflammatory diseases such as NS throughout life remains unprecedented.

ELIGIBILITY:
Inclusion Criteria:

Group A:

* Children aged 10 years and older and adults with confirmed Netherton syndrome diagnosed at age 10 years or older (clinical and histological and/or molecular)
* Patients and legal guardians informed about the study and not opposed to participation in the study

Group B:

* Children aged 10 years and older and adults with no skin barrier impairment, dermatosis, inflammatory disease, or autoimmune disease.
* Subjects and legal guardians informed about the study and who do not object to participation in the study.

Exclusion Criteria:

* Refusal by parents/guardians, children, adolescents, or adults.
* General or local antibiotic therapy within the month preceding the consultation.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion of children, adolescents, and young adults with Netherton syndrome, and control subjects of the same age and sex, treated at the service but without dermatosis or inflammatory and/or autoimmune diseases.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Study of the skin, salivary and intestinal microbiota | Baseline
  Analyse the skin microbiome, mycobiome, and virome, as well as the intestinal and salivary microbiome of patients with Netherton syndrome in comparison with healthy controls.

SECONDARY OUTCOMES:
Change in microbiome signature | Baseline
  Identify any changes in the microbiome signature of patients with Netherton syndrome.
Microbial interactions of the skin | Baseline
  Study the relationship between the different skin microbiome, mycobiome, and virome
Circulating cytokine profiles | Baseline
  Study circulating cytokine profiles
Markers of digestive inflammation | Baseline
  Study markers of digestive inflammation in stool samples
Factors influencing the microbiota | Baseline
  Analyze parameters that may impact the microbiotes, including various elements from these patients medical histories.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Necker Enfants Malades, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No